CLINICAL TRIAL: NCT04745585
Title: External Compression of the Abdominal Aorta to Reduce Femoral Arterial Flow: Comparison Between the Manual Technique and the New Echo-guided Technique
Brief Title: POCUS-PEAC to Reduce Femoral Arterial Blood Flow
Status: Terminated | Type: Observational
Why Stopped: Adverse event
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Raoul Daoust, Dr, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2020-1941
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the efficacy on healthy subjects of Point of Care ultrasonographically guided external aortic compression compared to the manual technique already described.

DETAILED DESCRIPTION:
Manual Proximal External Aortic Compression (M-PEAC) has been described for temporizing non-compressible hemorrhage. Point of Care Ultrasonographically guided External Aortic Compression (POCUS-PEAC), a new technique, has been used for management of junctional hemorrhage. The aim of this study is to compare the efficacy of US-PEAC to M-PEAC in reducing the distal arterial flow. This study also evaluates whether a small weight operator would benefit most of the US-PEAC compared to a standard weight operator. Other objectives are to evaluate pain and secondary effects. We will conduct an experimental crossover trial on healthy volunteers. Subjects will be recruited using a convenient sample. M-EAC and US-EAC will be performed on each subject. Femoral arterial flows will be measured by Doppler before and after each compression. Femoral flow reduction will be calculated for each technique and compared. The compression will be first accomplished by an 80 kg operator followed by a 57 kg operator. After each compression, pain will be evaluated using a visual analog scale (VAS). Fifteen minutes after the intervention, pain will be recorded using the same VAS. A follow-up will be ensured at 24 hours and at one week to evaluate for secondary effects.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 40 years old

Exclusion Criteria:

* <18 years old, >40 years old, BMI <18 or >25, History of abdominal surgery, history of vascular surgery, known aortic disease, known peripheral vascular disease, coronary disease, smoking, history of smoking, diabetes, dislipidemia, arterial hypertension, abdominal or inguinal hernia, eating in the last 4 hours before intervention, abdominal pain on the day of intervention, abdominal bloating on the day of intervention, pregnancy, impossibility to visualize the aorta with the ultrasound

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the flow reduction for each compression technique | 20 seconds
  For each subject, a nurse working at the vascular laboratory will measure the femoral arterial flow using Doppler ultrasound. A measurement will be noted before the interventions, after 20 seconds of manual compression, before the second intervention and after 20 seconds of POCUS compression. The reduction of flow will be calculated for each compression technique and the difference of reduction will be compared. The difference in flow reduction will also be compared for the small weight operator. The two operators will be blinded to the results.

SECONDARY OUTCOMES:
Subject pain evaluation | 15 minutes
  After each compression technique, the subject will be asked to evaluate the pain related to the intervention using a visual analogous scale (VAS)
  Fifteen minutes after the completion of the intervention, they will be asked to reposition their residual discomfort on the VAS.
Side effects | 7 days
  An assistant will call the subject at 24 hours following the intervention and at 7 days following the intervention to inquire about the presence of side effects (medical consultation, abdominal pain or other symptoms noted).

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Daoust, MD, MSc, Principal Investigator — Universite de Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada